CLINICAL TRIAL: NCT04987190
Title: Progressive Comparison of Density Assessment of Alveolar Bone Graft in Patients With Unilateral and Bilateral Cleft
Brief Title: Progression of Grafted Bone Density in Cleft Alveolus
Acronym: CDAABG
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pangyunchou, Craniofacial Research Center, Chang Gung Memorial Hospital
Other Study IDs: 201600968A3
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Cleft Lip and Palate
Keywords: alveolar bone grafting; alveolar cleft; bone mineral density; density enhancement rate; cone beam computed tomography (CBCT)
MeSH Terms: conditions — Cleft Lip | interventions — Alveolar Bone Grafting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all cleft patients divided into unilateral and bilateral groups: One group of cleft patients received the alveolar bone graft surgery
  Interventions: Procedure: alveolar bone graft

INTERVENTIONS:
Procedure: alveolar bone graft — alveolar bone graft with Scarpa fascia done when patients were at 9 year of age

SUMMARY:
The patients with unilateral and bilateral cleft lip and palate received alveolar bone graft surgery. Two time points of cone beam CT were taken for all the patients: post-operative 6 months, and post-operative 2 years. All the CT images were reviewed for the analysis of grafted bone density.

DETAILED DESCRIPTION:
Patient Information and Data Collection Patients who had nonsyndromic unilateral or bilateral cleft lip and alveolus with or without cleft palate and received ABG at our center between 2016 and 2018 were enrolled. All patients underwent at least 2 CBCT scans after operation. Postoperative image acquisition was performed at two time points, namely 6 months (T1) and 2 years (T2) after ABG. The ABG procedures for all patients were performed by the same senior surgeon per the protocol of our center, which comprises an iliac cancellous bone graft and the sealing of the Scarpa fascia to the defect before the bone graft is packed.2,12 Patient who had syndromic cleft alveolus, who underwent two-stage ABG (performed for bilateral cases), or who exhibited failed grafted tissue were excluded. In total, 40 patients were enrolled in the present study. The demographic and clinical variables for ABG were retrospectively collected through a review of medical charts. All CBCT images were obtained using an i-CAT CBCT scanner (Imaging Sciences International, Hatﬁeld, PA, USA); the parameters for the images are as follows: 120 kVp, voxel size of 0.4 × 0.4 × 0.4 mm3, 40-s scan time, and 22 × 16-cm field of view.

BMD Measurement The Picture Archiving and Communication System (PACS) was applied for image analysis. In addition, areas of interest were checked in the axial view slice by slice to locate the grafted tissue. Three methods (A, B, and C), which differed by the size of the selected area, were designed to measure Hounsfield units (HU). For all methods, we first identified the most superior and inferior planes transecting the grafted tissue. Subsequently, the middle plane of the grafted tissue was identified. For the selected plane, the distance between two teeth had to be larger than 2.5 mm in diameter; this was required for all three methods. On each plane, the selected circular area is defined as being located at the midpoint of the line between the centers of the two adjacent teeth. The HU of the selected area could be obtained using PACS.

For Method A, the circular zone located 1 mm from the adjacent teeth was selected. For Method B, the largest circular zone that exactly transected the two adjacent teeth or was tangent to the surrounding cortical bone was selected. For Method C, a circle was drawn with a diameter of 2 mm. Furthermore, an area of 2 × 0.5 mm2 in the pogonion was selected to obtain its HU at T1 and T2; this was the reference for calibration (Figure, Supplemental Digital Content 1). HU was the reference for BMD13 and represented the average density of the three planes. Calibrated BMD (BMDc, %) was defined using the following formula:

〖BMD〗_c (%)=〖HU〗_(selected zone)/〖HU〗_pogonion ×100.

Density enhancement rate (%) was calculated using the following formula:

Density enhancing rate (%)= (〖BMD〗_cT2-〖BMD〗_cT1)/〖BMD〗_cT1 ×100, where BMDcT2 is BMDc measured at T2, and BMDcT1 is the BMDc at T1. All the BMD and pogonion density data were measured by one examiner and repeated twice on different dates that were separated by a 3-month interval; the second round of measurements was conducted without reference to the first-round measurements. The average of the six sets of data (two measurements for each of the three planes) was used for the final statistical analysis.

Statistical Analysis In the descriptive analysis, continuous variables were summarized by means ± standard deviations. All variables were examined for normal distribution using the Shapiro-Wilk test. Student's t-test was performed to compare the means of continuous variables with normal distribution, and a chi-squared test or Fisher's exact test was used for categorical data. Furthermore, we performed analysis of variance with repeated measures to compare the differences between the three methods with respect to BMDc measurements and density enhancement rates in normally distributed data; for data that were not normally distributed, Friedman test was used. To compare the differences in BMDc at T1 and T2, we performed a paired t-test and a Wilcoxon signed-rank test for bilateral cleft due to small sample size. Bland-Altman plots were used to evaluate the agreement of each method. Intrarater reliability for the three methods was calculated using intraclass correlation coefficients (ICCs). All statistical tests were two-tailed, and a p value less than 0.05 was considered statistically significant. All data were analyzed using SPSS 24.0 (SPSS, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients who had nonsyndromic unilateral or bilateral cleft lip and alveolus with or without cleft palate
* Patients received alveolar bone graft at their 9 years of age
* Patients received twice CBCT after the surgery

Exclusion Criteria:

* Patient had syndromic cleft alveolus
* Patient underwent two-stage ABG (performed for bilateral cases)
* Patient exhibited failed grafted tissue

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In total, 40 patients, who had an average age of 9.45 ± 1.61 years when they received ABG, were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
mean calibrated bone mineral density (BMD/pogonion density, BMDc) | 1st BMD at post-operative 6 months
  BMD presented from CBCT
mean calibrated bone mineral density (BMD/pogonion density, BMDc) | 2nd BMD at post-operative 2 years
  BMD presented from CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Pangyun Chou, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan